CLINICAL TRIAL: NCT03599804
Title: Vestibular Function in Cochlear Implanted Hearing Impaired Children
Brief Title: Vestibular Cochlear Implant Hearing Impaired Child
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Hussein Ahmed Hamza, Principal investigator, Assiut University
Other Study IDs: VCIHIC
Record Dates: First submitted 2018-07-14; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Vestibular Abnormality
Keywords: Vestibular; Cochlear; Implant; Hearing; Child

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Cochlear implantation (CI) is a well-known surgical procedure to rehabilitate patients with severe to profound sensorineural hearing loss. Indications for this surgery have expanded in the last 10 years including bilateral CI. Although CI has been described as a safe procedure with few major complications, it may have an adverse effect on the vestibular functions and produce dizziness. Prevalence of postoperative dizziness varies widely in the literature and is said to affect between 2% - 47%.

DETAILED DESCRIPTION:
The structural and functional integrity of the vestibular system is necessary for maintenance of the complex postural system and adaptation to the environment. The absence of vestibular function is accompanied by poor prognosis and severe limitations in the activities of daily life, such as ambulating in low-light environments or on uneven ground, swimming, driving fast, etc.

The exact mechanisms responsible for the postoperative vestibular changes and/or symptoms, but several theories exist. Because of the very anatomic proximity between the auditory and vestibular systems, and their embryologic and physiologic alterations, they may be simultaneously involved in some bodily dysfunctions. This involvement is more frequent in peripheral alterations than in central ones.

The lateral wall and the fluid space are breached during cochleostomy. Insertion of electrode array may cause changes in the normal fluid homeostasis of the inner ear, damage to the basilar membrane, osseous spiral lamina and vestibular receptors; utricle, saccule and semicircular canals, surgery-induced inflammation resulting in fibrosis or loss of hair cells, foreign body reaction (labyrinthitis), produce perilymph leakage and alter the pressure in the inner ear. In addition, the electric stimulation of the cochlear implant may cause pathologic changes in the inner ear as a subsequent dysfunction of structures, resulting in vestibular alterations.

In previous research, the following vestibular assessments were utilized to determine vestibular injuries after CI: Caloric response, videonystagmography (VNG), vestibular-evoked myogenic potentials (VEMPs), video head impulse test (VHIT), rotatory chair and scleral search coil.

Knowledge of vestibular system function before and after CI surgery is important for the satisfactory management of each case. It also helps in the selection of which ear to implant to avoid bilateral vestibular areflexia and can assist in the management of any postoperative vestibular symptoms. So, there are two questions that should be raised when we consider the vestibular function of a patient who will submitted to CI: Is vestibular function present or not? and is the function symmetric?

ELIGIBILITY:
Inclusion Criteria:

1. Children with bilateral severe to profound sensorineural hearing loss.
2. Age less than 6years at time of implantation.
3. Prelingual deafness.

Exclusion Criteria:

* Incomplete follow up.
* Other pathologies affecting balance as orthopedic problems before surgery.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with severe to profound hearing loss aged less than 6 years and candidate for cochlear implant with no motor problems before surgery.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Head thrust test | baseline
  Clinical test which assesses vestibuloocular (VOR) function in which examiner briskly rotate patient's head to both sides while patient fixate his eyes on a target and watch for corrective saccades on eye movements.
Bruininks-Oseretsky test of motor proficiency (BOT-2) | baseline
  Clinical balance test which assesses vestibulospinal (VSR) function, patient stand on a firm surface and on a soft cushion with eyes closed and eye open, a scoring system is obtained for all these balance situations.
Caloric test | baseline
  Objective test of VOR, includes irrigation of warm and\or cool water into patient's external auditory canal and measure the resulting nystagmus by a computerized system.
Vestibular evoked myogenic potentials (VEMPs) | baseline
  Objective test of vestibulocollic (VCR) function which assesses otolithic organs, VEMPs amplitudes and latencies are measured by a computerized system.

CONTACTS AND LOCATIONS:
Overall Officials: Enass S Mohamed, MD, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bittar RSM, Sato ES, Ribeiro DJS, Tsuji RK. Preoperative vestibular assessment protocol of cochlear implant surgery: an analytical descriptive study. Braz J Otorhinolaryngol. 2017 Sep-Oct;83(5):530-535. doi: 10.1016/j.bjorl.2016.06.014. Epub 2016 Jul 31. PMID 27574724
- [Result] Krause E, Wechtenbruch J, Rader T, Gurkov R. Influence of cochlear implantation on sacculus function. Otolaryngol Head Neck Surg. 2009 Jan;140(1):108-113. doi: 10.1016/j.otohns.2008.10.008. PMID 19130972
- [Result] Todt I, Basta D, Ernst A. Does the surgical approach in cochlear implantation influence the occurrence of postoperative vertigo? Otolaryngol Head Neck Surg. 2008 Jan;138(1):8-12. doi: 10.1016/j.otohns.2007.09.003. PMID 18164986
- [Result] Kubo T, Yamamoto K, Iwaki T, Doi K, Tamura M. Different forms of dizziness occurring after cochlear implant. Eur Arch Otorhinolaryngol. 2001 Jan;258(1):9-12. doi: 10.1007/pl00007519. PMID 11271438
- [Result] Vibert D, Hausler R, Kompis M, Vischer M. Vestibular function in patients with cochlear implantation. Acta Otolaryngol Suppl. 2001;545:29-34. doi: 10.1080/000164801750388063. PMID 11677737
- [Result] Vibert D, Liard P, Hausler R. Bilateral idiopathic loss of peripheral vestibular function with normal hearing. Acta Otolaryngol. 1995 Sep;115(5):611-5. doi: 10.3109/00016489509139375. PMID 8928631
- [Result] Frazza MM. (1999): Propedèutica otoneurológica básica. In: Gananҫ, FF (coordenator). Um giro pela vertigem. Sào Paulo: Alaúde; p.21-24.
- [Result] Hempel JM, Jager L, Baumann U, Krause E, Rasp G. Labyrinth dysfunction 8 months after cochlear implantation: a case report. Otol Neurotol. 2004 Sep;25(5):727-9. doi: 10.1097/00129492-200409000-00014. PMID 15354003
- [Result] Katsiari E, Balatsouras DG, Sengas J, Riga M, Korres GS, Xenelis J. Influence of cochlear implantation on the vestibular function. Eur Arch Otorhinolaryngol. 2013 Feb;270(2):489-95. doi: 10.1007/s00405-012-1950-6. Epub 2012 Apr 6. PMID 22481544